CLINICAL TRIAL: NCT02283424
Title: A Randomized ,Opened, Prospective Controlled Trial of Clinical Effectiveness for Icotinib as the Adjunctive Treatment After Surgery in Stage I-IIIB Lung Adenocarcinoma Patients With Epidermal Growth Factor Receptor Gene Mutation
Brief Title: Icotinib as the Adjunctive Treatment After Surgery in Stage I-IIIB Lung Adenocarcinoma Patients With EGFR Gene Mutation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Liu, M.D., Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLATS1401
Record Dates: First submitted 2014-10-30; First posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Neoplasms, Therapy-Associated
MeSH Terms: conditions — Neoplasms, Second Primary | interventions — icotinib; Drug Therapy; Carboplatin; Docetaxel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemotherapy (Active Comparator): Carboplatin,350mg/m2,1/3weeks Docetaxel,75mg/m2,1/3weeks
  Interventions: Drug: Icotinib; Drug: chemotherapy (Carboplatin and Docetaxel)
- Icotinib (Experimental): Icotinib, 125mg,3/D,2years
  Interventions: Drug: Icotinib; Drug: chemotherapy (Carboplatin and Docetaxel)

INTERVENTIONS:
Drug: Icotinib — compared with chemotherapy,which is better for lung adenocarcinoma patients with epidermal growth factor receptor gene mutation after surgery
  Other Names: Conmana
Drug: chemotherapy (Carboplatin and Docetaxel) — as control group,compared with Icotinib
  Other Names: Carboplatin and Docetaxel

SUMMARY:
This is a randomized ,opened, prospective controlled trial of clinical effectiveness for Icotinib as the adjunctive treatment after surgery in stage I-IIIB lung adenocarcinoma patients with epidermal growth factor receptor gene mutation

DETAILED DESCRIPTION:
In this trial the investigators will enlist 100 patients who accepted surgery and with epidermal growth factor receptor gene mutation,these patients will be divided into 2 groups (chemotherapy group and Icotinib group),compare the PFS,RFS,OS after 5 years follow up

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Lung adenocarcinoma patients with epidermal growth factor receptor gene mutation,stage I-IIIB after surgery
* The patients' Eastern Cooperative Oncology Group scores are ≤ 0-2

Exclusion Criteria:

* Mismatch conditions above
* Have used other anti-cancer therapy drug before the trial and may influence the outcome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free Survival | 6 months

SECONDARY OUTCOMES:
Overall survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yang Liu, doctor, Study Chair — PLA General Hospital
Locations (1):
- PLA General Hospital, Beijing, China